CLINICAL TRIAL: NCT07317687
Title: Rapid HIV, Hepatitis C, and Syphilis Screening in a Rural Street Medicine Clinic in West Virginia
Brief Title: Rapid HIV, Hep C, and Syphilis Screening in a Rural Street Medicine Clinic
Status: Not yet recruiting | Type: Observational
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Madison Humerick, Assistant Professor, Department of Family Medicine - Eastern, West Virginia University
Other Study IDs: 2507193944
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: HIV Testing; HEPATITIS C (HCV); Syphilis; Hepatitis B Virus (HBV)
Keywords: Street Medicine; Rapid Fingerstick Testing
MeSH Terms: conditions — Hepatitis C; Syphilis; Hepatitis B | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Participants receiving fingerstick test: * Will get a quick fingerstick test for HIV, Hepatitis C, and syphilis.
  * Will receive results in 10-20 minutes.
  * If positive, will be offered immediate care and/or a referral.
  * If positive, blood draw will be offered on site to confirm results or referred to a WVU Medicine clinic location for follow-up blood test.
  * Will be invited to answer survey questions about the feelings and experiences with screening (about 15-30 minutes).
  Interventions: Diagnostic Test: Rapid Fingerstick Test
- Participants receiving blood-draw test: Participants receiving blood-draw test:
  * Will get a blood draw to test for HIV, Hepatitis B & C, and syphilis
  * Will receive results in approximately 3 days (via MyChart message and phone call, or in person at site)
  * If positive, will be offered immediate care and/or a referral for follow-up care. • Will be invited to answer questions about the feelings and experiences with screening (about 15 minutes).
  Interventions: Diagnostic Test: Blood Draw for lab test
- Participants who decline screening: Participants who decline screening:
  • Will be invited to answer survey questions about the feelings and experiences with screening (about 15-30 minutes).

INTERVENTIONS:
Diagnostic Test: Rapid Fingerstick Test — Fingerstick test for HIV, Hepatitis B and C, and Syphilis that gives results within 10-20 minutes
  Groups: Participants receiving fingerstick test
Diagnostic Test: Blood Draw for lab test — Blood draw to test for HIV, Hepatitis B & C, and syphilis which can take up to 3 days for results
  Groups: Participants receiving blood-draw test

SUMMARY:
West Virginia faces rising rates of HIV, hepatitis, and syphilis, particularly among individuals experiencing homelessness, substance use, and mental health challenges. Traditional blood-draw testing for these infections is often hindered by mistrust, logistical barriers, and delays in results. This study, conducted by the West Virginia University (WVU) Street Medicine program, evaluates a rapid, point-of-care fingerstick test for HIV, Hepatitis C, and syphilis that provides results within 10-20 minutes during mobile clinic visits. Participants may choose rapid testing, traditional blood draw (which also includes Hepatitis B screening), or decline testing. All participants will be invited to complete a brief survey about the experiences with screening methods. The goal is to assess whether rapid testing improves screening uptake, linkage to care, and patient satisfaction, ultimately reducing barriers and disease burden in high-risk populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the WVU Medicine Street Medicine team

Exclusion Criteria:

* Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will include patients in Berkeley and Jefferson Counties of West Virginia who visit the WVU Medicine Street Medicine Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Finger Stick | Day 1
  Percentage of participants that opted to take the rapid finger stick test.
Percentage of Blood Draw | Day 1
  Percentage of participants that opted to take the blood draw test.
Percentage that decline screening | Day 1
  Percentage of participants that opted to decline screening

CONTACTS AND LOCATIONS:
Overall Officials: Madison Humerick, MD, Principal Investigator — West Virginia University
Locations (1):
- WVU Department of Family Medicine - Eastern Division, Harpers Ferry, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No